CLINICAL TRIAL: NCT05860803
Title: Home-based, Digitally Delivered Breathing Training in People With Non-cystic Fibrosis Bronchiectasis: A Randomized Control Trial
Brief Title: Breathing Training and Exercise Capacity in Non-CFB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan Taylor, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-002736
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study staff who administer clinical testing before and after LT-PR will be blinded to the patient's group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control group of standard physician directed care (No Intervention): Subjects will receive pulmonary rehabilitation via standard physician directed care (i.e., 'normal care').
- Home-based specific breathing and respiratory muscle training group (Experimental): In addition standard of care pulmonary rehabilitation, subjects will participate in an 8-week home-based specific breathing and respiratory muscle training via the LungTrainers Pulmonary Rehabilitation regime (LT-PR).
  Interventions: Device: LungTrainers; Behavioral: LungTrainers Pulmonary Rehabilitation regime

INTERVENTIONS:
Device: LungTrainers — A training device that provides a variable resistance against which users breathe out. Users breathe through a plastic mouthpiece that is connected to an acrylic cylinder via rubber tubing. The mouthpiece has several small holes of various diameters and up to three stainless steel weights (half-weight increments) can be inserted into the acrylic tube. With each breath-out, the user exhales against the resistance provided by the weight inserts, and each inspiration (i.e., breath-in) is unresisted. During each resisted exhalation, the weight inserts are 'lifted' within the acrylic tube depending on the level of expiratory pressure generated by the participant.
  Arms: Home-based specific breathing and respiratory muscle training group
Behavioral: LungTrainers Pulmonary Rehabilitation regime — Series of different exercises using the LungTrainers device 3-5 days per week for approximately 10 weeks. Exercises complete in one long session (20-30 minutes) or be broken down into multiple shorter sessions (e.g., 3 x 10 minutes). A health coach will be assigned to guide participants through the LT-PR program.
  Other Names: LT-PR
  Arms: Home-based specific breathing and respiratory muscle training group

SUMMARY:
The purpose of this research is to investigate whether a home-based and health coach supported specific breathing and respiratory muscle training program improves the ability to exercise, the function of the lungs and breathing muscles, and general clinical status in people with non-cystic fibrosis bronchiectasis (non-CFB).

ELIGIBILITY:
Inclusion Criteria:

* Mayo Clinic patient with confirmed diagnosis of Non-Cystic Fibrosis Bronchiectasis (non-CFB): Non-CFB as confirmed by clinical history, including cough, shortness of breath, exertional dyspnea, pulmonary function tests, and high-resolution computed tomography. Patients will be considered clinically stable if there is no evidence of an exacerbation or change(s) in medical therapy in the previous three weeks.
* Able and willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Presence of significant coexisting disease, neurological conditions, and/or orthopedic complications that affect ability to undertake exercise.
* Presence of advanced heart failure.
* Current use of antibiotics.
* Acute exacerbation(s) within 3-weeks prior to study commencement.
* Participation within a pulmonary rehabilitation program within 6-months prior to study commencement.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in six-minute walk test distance | Baseline, 8 weeks
  Measures the distance walked in meters for 6 minutes.
Change in peak oxygen uptake during maximal incremental exercise test | Baseline, 8 weeks
  Maximum volume or amount of oxygen consumption during cardiopulmonary exercise test (treadmill or cycle).

SECONDARY OUTCOMES:
Change in exercise time during maximal incremental exercise test | Baseline, 8 weeks
  Maximum volume or amount of oxygen consumption during cardiopulmonary exercise test (treadmill or cycle).
Peak exercise work rate during maximal incremental exercise test | Baseline, 8 weeks
  Highest work rate achieved during cardiopulmonary exercise test (treadmill or cycle)
Change in forced vital capacity | Baseline, 8 weeks
  Measured by spirometry to determine the maximal amount of air that can be forcibly exhaled from the lungs after a full inhale, reported as liters (L).
Change in forced expiratory volume in 1 second | Baseline, 8 weeks
  Measured by spirometry to determine the volume of air that can be exhaled in 1 second with a forced breath.
Change in maximal voluntary ventilation | Baseline, 8 weeks
  Measured by spirometry to determine the largest amount of air inhaled and exhaled during maximal voluntary effort.
Change in maximal inspiratory pressure | Baseline, 8 weeks
  Assessed using a calibrated pressure meter to evaluate inspiratory muscle strength. After exhaling slowly and maximally (i.e., to residual volume), the subject will be urged strongly to 'suck-in as maximally as possible' (Mueller maneuver) for approximately 3 to 5 seconds. Measured by 3-5 repetitions and defined as the highest value (in cmH2O) of three measurements that vary by ≤5%.
Change in maximal expiratory mouth pressure | Baseline, 8 weeks
  Assessed using a calibrated pressure meter to evaluate expiratory muscle strength. After inhaling slowly and maximally (i.e., to total lung capacity), the patient will be strongly urged to 'blow-out as maximally as possible' (Valsalva maneuver) for approximately 3 to 5 seconds. Measured by 3-5 repetitions and defined as the highest value (in cmH2O) of three measurements that vary by ≤5%.
Change in diaphragm thickness | Baseline, 8 weeks
  Ultrasound-derived diaphragm thickness, reported centimeters (cm)
Change in diaphragm thickening fraction | Baseline, 8 weeks
  Ultrasound-derived diaphragm thickening fraction defined as ratio of at total lung capacity thickness at functional residual capacity to thickness at functional residual capacity, reported in millimeters (mm).
Change in diaphragm excursion | Baseline, 8 weeks
  Ultrasound-derived diaphragm excursion defined as the amplitude of excursion from baseline to the point of maximum height during the sniff, reported in centimeters (cm).
Change in Modified Medical Research Council Dyspnea Scale (mMRC) | Baseline, 8 weeks
  mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4 which 0=no breathlessness except on strenuous exercise; 1=shortness of breath when hurrying on the level or walking up a slight hill; 2=walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3=stops for breath after walking approximately 100 m or after few minutes on the level; and 4=too breathless to leave the house, or breathless when dressing or undressing.
Change in St. George's Respiratory Questionnaire (SGRQ) | Baseline, 8 weeks
  SGRQ measures impact on overall health, daily life, and perceived well-being in patients with lung disease, specifically obstructive airways disease. The questionnaire consists of two parts with three components; Part 1: symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall. Scores range from 0 to 100, with higher scores indicating more limitations.
Change in Dartmouth COOP Functional Assessment Charts | Baseline, 8 weeks
  The Dartmouth COOP chart consists of nine questions measuring seven domains of health status: physical fitness, feelings, daily activities, social activities, change in health status, current overall health perceptions, bodily pain, social support, and quality of life. Each question has five response options.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Taylor, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials